CLINICAL TRIAL: NCT01145079
Title: A New Strategy Regarding Discontinuation of Dual Antiplatelet; Real Safety and Efficacy of a 3-month Dual Antiplatelet Therapy Following Zotarolimus-eluting Stents Implantation (RESET Trial)
Brief Title: A New Strategy Regarding Discontinuation of Dual Antiplatelet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2009-0115
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Endeavor arm (Experimental)
  Interventions: Device: Zotarolimus-eluting stent
- Endeavor resolute arm (Active Comparator)
  Interventions: Device: Zotarolimus-eluting stent for ACS and DM
- Xience arm (Active Comparator)
  Interventions: Device: Everolimus-eluting stent for long lesion
- Cypher arm (Active Comparator)
  Interventions: Device: Sirolimus-eluting stent for short lesion

INTERVENTIONS:
Device: Zotarolimus-eluting stent — Zotarolimus-eluting stent
  Arms: Endeavor arm
Device: Zotarolimus-eluting stent for ACS and DM — Zotarolimus-eluting stent for ACS and DM
  Arms: Endeavor resolute arm
Device: Everolimus-eluting stent for long lesion — Everolimus-eluting stent for long lesion
  Arms: Xience arm
Device: Sirolimus-eluting stent for short lesion — Sirolimus-eluting stent for short lesion
  Arms: Cypher arm

SUMMARY:
Drug-eluting stents (DES), markedly reducing the neointimal hyperplasia after stent implantation compared with bare-metal stents (BMS), have improved angiographic and clinical outcomes in the complex lesions and patients with high risks. However, currently, the fatal events related with stent thrombosis still occur and are the major limitation of the use of DES. Especially, late or very late thrombosis after DES implantation is an uncommon but life-threatening fatal complication presented with sudden death or myocardial infarction (MI) causing heart failure. The most powerful predictor for stent thrombosis is the discontinuation of clopidogrel. In consideration of current data regarding stent thrombosis and clinical situation of discontinuation of antiplatelet, zotarolimus-eluting stent (ZES) [Endeavor®, Medtronic Vascular, Santa Rosa, CA] might be anticipated to be safer than other DES during the long-term follow-up owing to healthy endothelialization. Endeavor® stent was consists of zotarolimus, thin-strut, cobalt-chromium alloy stent platform (DriverTM stent; Medtronic Vascular, Santa Rosa, CA), and phosphorylcholine coating. The ENDEAVOR II study demonstrated clinically and statistically significant improvement in all of study endpoints, including a 47 percent reduction in the primary endpoint of target vessel failure (TVF). In addition, the ENDEAVOR II trial showed a 0.5 percent rate of stent thrombosis at 30 days - with no late thrombosis beyond 30 days and no late stent malapposition. Because reendothelialization after ZES implantation may occur within 3 months, 3-month dual antiplatelet therapy is recommended in many clinical trials and real world practice. Shorter maintenance of dual antiplatelet therapy might minimize the risk for stent thrombosis in cases of discontinuation of antiplatelet and prevent waste medications and bleeding complications related with dual antiplatelet therapy. However, there have been no non-inferior or superior data of ZES considering all these circumstances. Therefore, the investigators hypothesize that ZES with 3-month dual antiplatelet therapy may be safe and beneficial in patients with coronary artery disease during follow-up than other DES, in spite of higher late lumen loss. To test this hypothesis, the investigators will perform a multi-center, randomized, prospective trial aimed at demonstrating the efficacy of the ZES versus other DES in patients with coronary artery disease in real world practice.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease including stable angina, unstable angina, acute non-ST elevation myocardial infarction and acute ST elevation myocardial infarction
* Age 20 years of older
* Patients with typical chest pain or evidences of myocardial ischemia (e.g., stable, unstable angina, silent ischemia and positive functional study or reversible changes in the electrocardiogram (ECG) consistent with ischemia
* Patients with signed informed consent
* Lesion and stent length for ACS and DM subgroup : Length of single lesion < 24 mm and, Summation of total length of all inserted DES in 3 vessel < 60 mm
* Lesion and stent length for ACS and DM subgroup : Length of single lesion < 24 mm and, Summation of total length of all inserted DES in 3 vessel < 60 mm
* Lesion and stent length for long lesion subgroup : Length of single stent per single lesion > 28 mm and, Summation of total length of all inserted DES in 3 vessel ≤ 90 mm, Possible overlapping stent
* Lesion and stent length for short lesion subgroup : Length of single lesion < 24 mm and, Summation of total length of all inserted DES in 3 vessel < 60 mm
* Significant coronary artery stenosis (>50% by visual estimate) considered for coronary revascularization with stent implantation
* Reference vessel diameter of 2.5 to 4.0 mm by operator assessment
* Lesion success (30% or less residual stenosis by visual assessment over the entire stent length, with TIMI-3 flow and no more than an NHLBI type B peri-stent dissection

Exclusion Criteria:

* Contraindication to anti-platelet agents & bleeding history within prior 3 months
* Known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, limus related drug
* Prior history of the following presentations : Cerebral vascular accident (not including transient ischemic attack, Peripheral artery occlusive diseases, Thromboembolic disease, Stent thrombosis
* Severe hepatic dysfunction (3 times normal reference values)
* Significant renal dysfunction (Serum creatinine > 2.0 mg/dl)
* Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
* Cardiogenic shock
* LVEF < 40%
* Pregnant women or women with potential childbearing
* Life expectancy 3 year
* Overlapped DESs(only long lesion subgroup is possible overlapping)
* Left main disease requiring PCI
* Bifurcation lesion with 2-stent technique
* Target lesions with in-stent restenosis at the stented segment of DES or BMS
* Lesions with chronic total occlusion
* History of PCI with DES
* In-stent restenosis lesion

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 982 (Actual)
Dates: Start 2009-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome The composite of cardio-vascular death, MI, stent thrombosis, TVR and bleeding (minor or major) following randomly assigned DES implantation | 12 months after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Myeong Ki Hong, MD, PhD, Principal Investigator — Severance Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Jin IT, Kim Y, Heo SJ, Lee YJ, Lee SJ, Hong SJ, Ahn CM, Kim JS, Cho DK, Ko YG, Choi D, Hong MK, Kim BK. Comparison of Short-term and Standard Duration Dual Antiplatelet Therapy in Elderly Patients: A Pooled Analysis of Five Korean Randomized Clinical Trials. Korean Circ J. 2025 Dec;55(12):1125-1137. doi: 10.4070/kcj.2025.0093. Epub 2025 Jul 14. PMID 41044734
- [Derived] Jang JY, Jung HW, Lee BK, Shin DH, Kim JS, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Park KW, Gwon HC, Kim HS, Kwon HM, Jang Y. Impact of PRECISE-DAPT and DAPT Scores on Dual Antiplatelet Therapy Duration After 2nd Generation Drug-Eluting Stent Implantation. Cardiovasc Drugs Ther. 2021 Apr;35(2):343-352. doi: 10.1007/s10557-020-07008-7. PMID 32588238
- [Derived] Jang JY, Shin DH, Kim JS, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Park KW, Gwon HC, Kim HS, Jang Y. Optimal duration of DAPT after second-generation drug-eluting stent in acute coronary syndrome. PLoS One. 2018 Nov 26;13(11):e0207386. doi: 10.1371/journal.pone.0207386. eCollection 2018. PMID 30475845
- [Derived] Kim JS, Kang TS, Mintz GS, Park BE, Shin DH, Kim BK, Ko YG, Choi D, Jang Y, Hong MK. Randomized comparison of clinical outcomes between intravascular ultrasound and angiography-guided drug-eluting stent implantation for long coronary artery stenoses. JACC Cardiovasc Interv. 2013 Apr;6(4):369-76. doi: 10.1016/j.jcin.2012.11.009. Epub 2013 Mar 20. PMID 23523455
- [Derived] Kim BK, Hong MK, Shin DH, Nam CM, Kim JS, Ko YG, Choi D, Kang TS, Park BE, Kang WC, Lee SH, Yoon JH, Hong BK, Kwon HM, Jang Y; RESET Investigators. A new strategy for discontinuation of dual antiplatelet therapy: the RESET Trial (REal Safety and Efficacy of 3-month dual antiplatelet Therapy following Endeavor zotarolimus-eluting stent implantation). J Am Coll Cardiol. 2012 Oct 9;60(15):1340-8. doi: 10.1016/j.jacc.2012.06.043. Epub 2012 Sep 19. PMID 22999717